CLINICAL TRIAL: NCT01972308
Title: A Patient Advocate to Improve Real-world Asthma Management for Inner City Adults
Acronym: HAP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Andrea Apter, Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R18HL116285-01 (NIH)
Record Dates: First submitted 2013-10-16; First posted 2013-10-30 (Estimated); Results first posted 2018-08-06 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Asthma; Communication
Keywords: asthma; patient advocate; health disparity; patient-provider communication
MeSH Terms: conditions — Asthma; Communication

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient advocate (Experimental): Subject works with a Patient Advocate who coaches, models, and assists with preparations for a visit with the asthma doctor; attends the visit with permission of participant and provider; and confirms understanding. The PA facilitates scheduling, obtaining insurance coverage, overcoming patients' unique social and administrative barriers to carrying out medical advice, and transfer of information between providers and patients.
  Interventions: Behavioral: Patient Advocate
- usual care (Other): Patient receives asthma care as usual from their asthma provider
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Patient Advocate — Subject works with a Patient Advocate who coaches, models, and assists with preparations for a visit with the asthma doctor; attends the visit with permission of participant and provider; and confirms understanding. The PA facilitates scheduling, obtaining insurance coverage, overcoming patients' unique social and administrative barriers to accomplishing medical advice, and transfer of information between provider and patient.
  Arms: Patient advocate
Behavioral: Usual Care — Subjects receive asthma care from their proivders in the participating practices which generally follow asthma guidelines
  Arms: usual care

SUMMARY:
Few interventions to improve asthma management have targeted low-income minority asthmatic adults and even fewer have focused on the real-world practice where care is provided for these patients. This project tests the effectiveness of a Patient Advocate as a practical and sustainable method of facilitating and maintaining communication between patient and provider and access to chronic care for adults with moderate or severe asthma recruited from clinics serving low-income urban neighborhoods. We compare the use of a Patient Advocate to current asthma care and test the Patient Advocate's cost-effectiveness.

DETAILED DESCRIPTION:
This 5 year project tests the effectiveness, sustainability, and budget impact of a patient navigator intervention to facilitate and maintain patient-provider communication and access to chronic care of moderate or severe asthma in low income minority adults with other chronic morbidities. We will recruit from a variety of clinic practices including those of an urban academic health center, a VA, and a federally qualified health center and in both English-speaking and Spanish-speaking patients. The intervention is tailored to patients and their clinics, and informed by focus groups of patients and providers.

The Patient Advocate (PA), works with patients by coaching and modeling preparation for a visit with the asthma doctor, attending the visit with the permission of participant and provider, and confirming understanding of issues discussed. The PA also facilitates scheduling, obtaining insurance coverage, overcoming patients' unique social and administrative barriers to carrying out medical advice, and exchange of information between providers and patients. The PAs are recent college graduates interested in health-related or education careers, research experience, working with patients, and generally have the same race/ethnicity distribution as potential subjects.

This dissemination and implementation project refines the intervention of RC1 HL099612 for real-world practice by 1) conducting a randomized controlled trial that compares the Patient Advocate Intervention (PAI) to currently practiced guideline-based usual care; 2) carrying out the intervention in a variety of primary care and asthma specialty practices; 3) extending the observation time to a year to test its sustainability; 4) assessing patient-centered outcomes including asthma control, quality of life, ED visits, and hospitalizations; 5) assessing mediators/moderators of the PAI-asthma outcome relationship; and 6) evaluating its cost-effectiveness.

We will recruit 300 adults, each to be followed for at least 1 year with moderate or severe persistent asthma from clinics serving low-income, urban, primarily minority patients and conduct a randomized controlled trial (RCT) to: 1) assess whether 6 months of the PAI improves asthma control relative to baseline compared with usual care (UC) and whether such a difference is sustained in the 6 months following the intervention's completion, 2) Assess whether the PAI improves other asthma outcomes (need for prednisone bursts, ED visits, hospitalizations, quality of life, FEV1) relative to baseline compared with UC at 6 months and is sustained in the 6 months following the intervention's completion, 3) examine mediators and moderators of the relationship between the intervention and outcome, 4) assess the incremental direct and indirect costs of the PAI compared to usual care and the cost-effectiveness of the PAI relative to UC for the outcomes, and 5) in post-study focus groups of providers to explore awareness of the intervention and response to the PA

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age,
2. physician's diagnosis of asthma,
3. prescribed an inhaled-steroid-containing medication for asthma (ensuring the patient is believed to have moderate or severe reversible airways obstruction by their physician),
4. moderate or severe persistent asthma according to the NHLBI Guidelines,
5. evidence of reversible airflow obstruction: (a) forced expiratory volume in 1 second (FEV1) < 80% predicted at the time of screening or within the 3 years prior to this screening, and (b) improvement with bronchodilator: either (i) an increase of >15% and 200ml in FEV1 with asthma treatment over the previous 3 years or (ii) after 4 puffs of albuterol by MDI (or 2.5 mg by nebulizer), an increase in FEV1 or FVC >12% and 200 ml in FEV1 within 30 minutes,
6. at least one appointment scheduled with the asthma physician during the 1st 6 months of participation

Exclusion Criteria:

1. Severe psychiatric or cognitive problems (e.g., obvious mania, schizophrenia, significant mental retardation) that make it impossible to understand and carryout PA activities.
2. Unable to understand and provide informed consent,
3. Unable to communicate in English or Spanish.
4. Participants of the pilot study for this project are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2013-12-12 (Actual); Primary Completion 2017-03-16 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea J Apter, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Apter AJ, Wan F, Reisine S, Bogen DK, Rand C, Bender B, Bennett IM, Gonzalez R, Priolo C, Sonnad SS, Bryant-Stephens T, Ferguson M, Boyd RC, Ten Have T, Roy J. Feasibility, acceptability and preliminary effectiveness of patient advocates for improving asthma outcomes in adults. J Asthma. 2013 Oct;50(8):850-60. doi: 10.3109/02770903.2013.812655. Epub 2013 Jul 17. PMID 23800333
- [Background] Apter AJ, Wan F, Reisine S, Bender B, Rand C, Bogen DK, Bennett IM, Bryant-Stephens T, Roy J, Gonzalez R, Priolo C, Have TT, Morales KH. The association of health literacy with adherence and outcomes in moderate-severe asthma. J Allergy Clin Immunol. 2013 Aug;132(2):321-7. doi: 10.1016/j.jaci.2013.02.014. Epub 2013 Apr 13. PMID 23591273
- [Background] Apter AJ, Bryant-Stephens T, Morales KH, Wan F, Hardy S, Reed-Wells S, Dominguez M, Gonzalez R, Mak N, Nardi A, Park H, Howell JT, Localio R. Using IT to improve access, communication, and asthma in African American and Hispanic/Latino Adults: Rationale, design, and methods of a randomized controlled trial. Contemp Clin Trials. 2015 Sep;44:119-128. doi: 10.1016/j.cct.2015.08.001. Epub 2015 Aug 8. PMID 26264737
- [Background] Bryant-Stephens T, Reed-Wells S, Canales M, Perez L, Rogers M, Localio AR, Apter AJ. Home visits are needed to address asthma health disparities in adults. J Allergy Clin Immunol. 2016 Dec;138(6):1526-1530. doi: 10.1016/j.jaci.2016.10.006. Epub 2016 Oct 21. PMID 27777181
- [Background] Kramer CB, LeRoy L, Donahue S, Apter AJ, Bryant-Stephens T, Elder JP, Hamilton WJ, Krishnan JA, Shelef DQ, Stout JW, Sumino K, Teach SJ, Federman AD. Enrolling African-American and Latino patients with asthma in comparative effectiveness research: Lessons learned from 8 patient-centered studies. J Allergy Clin Immunol. 2016 Dec;138(6):1600-1607. doi: 10.1016/j.jaci.2016.10.011. Epub 2016 Oct 24. PMID 27789250
- [Background] Apter AJ, Perez L, Han X, Ndicu G, Localio A, Park H, Mullen AN, Klusaritz H, Rogers M, Cidav Z, Bryant-Stephens T, Bender BG, Reisine ST, Morales KH. Patient Advocates for Low-Income Adults with Moderate to Severe Asthma: A Randomized Clinical Trial. J Allergy Clin Immunol Pract. 2020 Nov-Dec;8(10):3466-3473.e11. doi: 10.1016/j.jaip.2020.06.058. Epub 2020 Jul 14. PMID 32673877
- [Background] Korwin A, Black H, Perez L, Morales KH, Klusaritz H, Han X, Huang J, Rogers M, Ndicu G, Apter AJ. Exploring Patient Engagement: A Qualitative Analysis of Low-Income Urban Participants in Asthma Research. J Allergy Clin Immunol Pract. 2017 Nov-Dec;5(6):1625-1631.e2. doi: 10.1016/j.jaip.2017.03.022. Epub 2017 May 10. PMID 28499772
- [Derived] Buckey TM, Morales KH, Apter AJ. Understanding Autonomy in Patients with Moderate to Severe Asthma. J Allergy Clin Immunol Pract. 2022 Feb;10(2):525-533. doi: 10.1016/j.jaip.2021.10.068. Epub 2021 Nov 14. PMID 34785390

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient Advocate: Subject works with a Patient Advocate who coaches, models, and assists with preparations for a visit with the asthma doctor; attends the visit with permission of participant and provider; and confirms understanding. The PA facilitates scheduling, obtaining insurance coverage, overcoming patients' unique social and administrative barriers to carrying out medical advice, and transfer of information between providers and patients.
  Patient Advocate: Subject works with a Patient Advocate who coaches, models, and assists with preparations for a visit with the asthma doctor; attends the visit with permission of participant and provider; and confirms understanding. The PA facilitates scheduling, obtaining insurance coverage, overcoming patients' unique social and administrative barriers to carrying out medical advice, and transfer of information between providers and patients
Period: Overall Study
Arm/Group | Patient Advocate | Usual Care
Started | 156 | 156
Completed | 148 | 148
Not Completed | 8 | 8
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 4 | 6
Not completed — Death | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Advocate | Usual Care | Total
Number analyzed (Participants) | 156 | 156 | 312
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (14.3) | 49.6 (13.7) | 51.1 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 115 | 216
  Male | 55 | 41 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 11 | 25
  Not Hispanic or Latino | 142 | 145 | 287
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 100 | 106 | 206
  White | 40 | 35 | 75
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 14 | 12 | 26
asthma control questionnaire [Mean (Standard Deviation); unit: units on a scale] — Asthma Control range is 0-6 with lower score better control (0= total control and 6 = extremetly uncontrolled. The minimally important clinical difference is 0.5. A score > 1.5 is considered inadequate control.
  units on a scale | 2.3 (1.1) | 2.4 (1.2) | 2.4 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Asthma Control at One Year
Description: Asthma Control Questionnaire: In a randomized controlled trial we will assess whether 6 months of the Patient Advocate Intervention improves asthma control relative to baseline compared with usual care (UC) and whether such a difference is sustained in the 6 months following the intervention's completion.
  Asthma Control range is 0-6 with lower score better control (0= total control and 6 = extremetly uncontrolled. The minimally important clinical difference is 0.5. A score > 1.5 is considered inadequate control.
Time Frame: baseline and 1 year
Population: 18 years or more, physician's diagnosis of asthma, prescribed an inhaled-steroid for asthma, moderate or severe persistent asthma, evidence of reversible airflow obstruction, at least one appointment scheduled with the asthma physician during the 1st 6 months of participation
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Patient Advocate | Usual Care
Number analyzed (Participants) | 156 | 156
units on a scale | -0.42 [-0.65 to -0.18] | -0.11 [-0.37 to 0.12]
Statistical Analysis 1: Comparison: Patient Advocate vs Usual Care; Test type: Superiority; Group differences in expected 12 month c = -0.31, 95% CI 2-sided [-0.64 to 0.04]

2. Secondary Outcome: Change in Emergency Department(ED) Visits at One Year
Description: Emergency room visits in the 6 months before entry compared with emergency room visits in the 6 months prior to the one year timepoint
Time Frame: one year
Measure: Least Squares Mean (95% Confidence Interval); unit: visits per 6 months
Arm/Group | Patient Advocate | Usual Care
Number analyzed (Participants) | 156 | 156
visits per 6 months | -0.90 [-1.50 to -0.42] | -0.24 [-0.60 to 0.18]
Statistical Analysis 1: Comparison: Patient Advocate vs Usual Care; Test type: Superiority; Group differences in expected 12 month c = -0.66, 95% CI 2-sided [-1.38 to -0.01]

3. Secondary Outcome: Change in Asthma-related Quality of Life
Description: Asthma-related quality of life will be measured with the Mini-Asthma Quality of Life Questionnaire (AQLQ). This 15-item questionnaire with each item having a 7-point response scale that provides a mean summary score. A 0.5-unit change is considered clinically meaningful. the range is 1 - 7 with higher score better quality of life.
Time Frame: baseline to one year
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Patient Advocate | Usual Care
Number analyzed (Participants) | 156 | 156
units on a scale | 0.28 [0.01 to 0.54] | 0.23 [-0.05 to 0.48]
Statistical Analysis 1: Comparison: Patient Advocate vs Usual Care; Test type: Superiority; Group differences in expected 12 month c = 0.06, 95% CI 2-sided [-0.33 to 0.43]

4. Secondary Outcome: Change in Hospitalizations
Description: Participants will report hospitalizations verified if possible in participating health systems. We review records and if not available ask patient for hospititalizations over the 6 months before baseline and compare it with the record or report in the 6-months prior to one year.
Time Frame: one year
Measure: Least Squares Mean (95% Confidence Interval); unit: hospitalizations per 6 months
Groups:
- Usual Care: Patient receives asthma care as usual from their asthma provider
  Patient Advocate: Subject works with a Patient Advocate who coaches, models, and assists with preparations for a visit with the asthma doctor; attends the visit with permission of participant and provider; and confirms understanding. The PA facilitates scheduling, obtaining insurance coverage, overcoming patients' unique social and administrative barriers to carrying out medical advice, and transfer of information between providers and patients
Arm/Group | Patient Advocate | Usual Care
Number analyzed (Participants) | 156 | 156
hospitalizations per 6 months | -0.30 [-0.66 to -0.06] | -0.36 [-0.66 to -0.12]
Statistical Analysis 1: Comparison: Patient Advocate vs Usual Care; Test type: Superiority; Group differences in expected 12 month c = 0.02, 95% CI 2-sided [-0.42 to 0.48]

5. Secondary Outcome: Risk of Prednisone Bursts
Description: a new dose or an increase in already prescribed prednisone dose
Time Frame: baseline and one year
Measure: Least Squares Mean (95% Confidence Interval); unit: risk of prednisone bursts
Arm/Group | Patient Advocate | Usual Care
Number analyzed (Participants) | 156 | 156
risk of prednisone bursts | -0.005 [-0.10 to 0.10] | -0.05 [-0.14 to 0.05]
Statistical Analysis 1: Comparison: Patient Advocate vs Usual Care; Test type: Superiority; Group differences in expected 12 month c = 0.04, 95% CI 2-sided [-0.10 to 0.19]

6. Secondary Outcome: Change in Urgent Office Visit
Description: Records or if not available patient report of an urgent office visit in the 6 months before baseline compared with record or report of urgent office visits in the 6 months prior to one year. An urgent office visit is one scheduled within 24 hours of the visit.
Time Frame: one year
Measure: Least Squares Mean (95% Confidence Interval); unit: urgent visits per 6 months
Arm/Group | Patient Advocate | Usual Care
Number analyzed (Participants) | 156 | 156
urgent visits per 6 months | -0.24 [-0.54 to 0.02] | -0.42 [-0.72 to -0.12]
Statistical Analysis 1: Comparison: Patient Advocate vs Usual Care; Test type: Superiority; Group differences in expected 12 month c = 0.12, 95% CI 2-sided [-0.24 to 0.60]

ADVERSE EVENTS:
Time Frame: one year
Arm/Group | Patient Advocate | Usual Care
All-Cause Mortality (participants affected / at risk) | 4/156 | 1/156
Serious Adverse Events (participants affected / at risk) | 89/156 | 90/156
Other Adverse Events (participants affected / at risk) | 71/156 | 74/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patient Advocate (N=156) | Usual Care (N=156)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 43 | 44
foot pain (Musculoskeletal and connective tissue disorders) | 5 | 2
short of breath (Respiratory, thoracic and mediastinal disorders) | 6 | 3
surgical and medical procedure (Surgical and medical procedures) | 14 | 7
abdominal pain (Gastrointestinal disorders) | 6 | 7
back pain (Musculoskeletal and connective tissue disorders) | 4 | 9
chest pain (Cardiac disorders) | 6 | 6
allergic reaction (Immune system disorders) | 4 | 4
fall (Injury, poisoning and procedural complications) | 3 | 5
ankle sprain (Injury, poisoning and procedural complications) | 3 | 5
skin abscess (Skin and subcutaneous tissue disorders) | 3 | 4
skin infection (Infections and infestations) | 4 | 3
urinary tract infection (Infections and infestations) | 3 | 4
headache (Nervous system disorders) | 2 | 5
injury, poisoning and procedural complication (Injury, poisoning and procedural complications) | 4 | 2
hypertension (Cardiac disorders) | 4 | 2
pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 | 3
acute sinusitis (Infections and infestations) | 3 | 3
upper respiratory infection (Infections and infestations) | 1 | 5
vomiting (Gastrointestinal disorders) | 4 | 2
sore throat (Respiratory, thoracic and mediastinal disorders) | 3 | 2
stomach pain (Gastrointestinal disorders) | 2 | 3
arthritis (Musculoskeletal and connective tissue disorders) | 1 | 3
constipation (Gastrointestinal disorders) | 2 | 2
hyperglycemia (Endocrine disorders) | 2 | 2
psychiatric disorder (Psychiatric disorders) | 3 | 1
skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 | 2
diverticulitis (Gastrointestinal disorders) | 2 | 1
hypoglycemia (Endocrine disorders) | 2 | 1
pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 3
bronchial infection (Infections and infestations) | 1 | 2
anxiety (Psychiatric disorders) | 1 | 1
chest wall pain (Cardiac disorders) | 1 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
flu-like symptoms (General disorders) | 0 | 2
fracture (Injury, poisoning and procedural complications) | 1 | 1
gastrointestinal disorders (Gastrointestinal disorders) | 1 | 1
acute and chronic respiratory failure with hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
respiratory, thoracic and medistinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 1
seizure (Nervous system disorders) | 1 | 1
skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
vaginal bleeding (Reproductive system and breast disorders) | 2 | 0
wheeze (Respiratory, thoracic and mediastinal disorders) | 0 | 2
lung infection (Infections and infestations) | 1 | 1
noncardiac chest pain (General disorders) | 0 | 2
GERD (Gastrointestinal disorders) | 1 | 1
anaphylaxis (Immune system disorders) | 1 | 0
anemia (Blood and lymphatic system disorders) | 1 | 0
ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 | 0
blurred vision (Eye disorders) | 1 | 0
bruising (Injury, poisoning and procedural complications) | 1 | 0
colitis (Gastrointestinal disorders) | 0 | 1
conjunctivitis (Eye disorders) | 0 | 1
dehydration (Metabolism and nutrition disorders) | 0 | 1
dental caries (Gastrointestinal disorders) | 1 | 0
depression (Psychiatric disorders) | 1 | 0
diarrhea (Gastrointestinal disorders) | 0 | 1
dry mouth (Gastrointestinal disorders) | 0 | 1
ear pain (Ear and labyrinth disorders) | 0 | 1
corneal abrasion (Eye disorders) | 0 | 1
eye irritation (Eye disorders) | 0 | 1
facial pain (Injury, poisoning and procedural complications) | 0 | 1
fatigue (General disorders) | 0 | 1
fever (General disorders) | 1 | 0
gait disturbance (General disorders) | 1 | 0
gall bladder pain (Gastrointestinal disorders) | 1 | 0
general disorders (General disorders) | 1 | 0
hematuria (Renal and urinary disorders) | 0 | 1
immune system disorders (Immune system disorders) | 1 | 0
knee swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 | 0
musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 | 1
trigeminal neurlagia (Nervous system disorders) | 1 | 0
ear infection (Infections and infestations) | 0 | 1
shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 1
palpitations (Cardiac disorders) | 1 | 0
paresthesia (Nervous system disorders) | 0 | 1
pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
pruritis (Skin and subcutaneous tissue disorders) | 0 | 1
kidney stone (Renal and urinary disorders) | 0 | 1
reproductive system and breast disorders (Reproductive system and breast disorders) | 1 | 0
sepsis (Infections and infestations) | 0 | 1
seroma (Injury, poisoning and procedural complications) | 1 | 0
sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
small intestine obstruction (Gastrointestinal disorders) | 0 | 1
stroke symptoms (Nervous system disorders) | 0 | 1
suicidal ideation (Psychiatric disorders) | 1 | 0
transient ischemic attack (Nervous system disorders) | 1 | 0
urinary retention (Renal and urinary disorders) | 0 | 1
uterine pain (Reproductive system and breast disorders) | 1 | 0
vaginal infection (Infections and infestations) | 0 | 1
deep venous thrombosis (Vascular disorders) | 0 | 1
ventricular arrhrythmia (Cardiac disorders) | 0 | 1
ear and labyrinth disorders (Ear and labyrinth disorders) | 1 | 0
corneal ulcer (Eye disorders) | 0 | 1
infection and infestations (Infections and infestations) | 0 | 1
edema (General disorders) | 1 | 0
angina (Cardiac disorders) | 1 | 0
peritoneal infection (Infections and infestations) | 0 | 1
sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
soft tissue infection (Infections and infestations) | 1 | 0
vulvovaginal candidiasis (Infections and infestations) | 1 | 0
foot weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patient Advocate (N=156) | Usual Care (N=156)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 29 | 31
short of breath (Respiratory, thoracic and mediastinal disorders) | 7 | 6
foot pain (General disorders) | 8 | 4
depression (Psychiatric disorders) | 4 | 4
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 6 | 2
headache (Nervous system disorders) | 2 | 5
sinusitis (Infections and infestations) | 4 | 3
skin disorders (Skin and subcutaneous tissue disorders) | 6 | 1
surgical and medical procedures (Surgical and medical procedures) | 3 | 3
abdominal pain (Gastrointestinal disorders) | 2 | 3
back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
chest pain (Cardiac disorders) | 2 | 3
cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
flu-like symptoms (General disorders) | 3 | 2
allergic reaction (Immune system disorders) | 2 | 2
fall (Injury, poisoning and procedural complications) | 1 | 3
abscess (Skin and subcutaneous tissue disorders) | 1 | 3
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 3
bronchial infection (Infections and infestations) | 3 | 1
arthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
hypertension (Cardiac disorders) | 3 | 0
neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1
arthralgia shoulder (Musculoskeletal and connective tissue disorders) | 2 | 0
gastrointestinal disorder (Gastrointestinal disorders) | 1 | 1
musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 | 1
neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
ear infection (Infections and infestations) | 2 | 0
pain (General disorders) | 1 | 1
cellulitis (Skin and subcutaneous tissue disorders) | 2 | 0
palpitations (Cardiac disorders) | 2 | 0
respiratory, thoracic, and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 1
skin infection (Infections and infestations) | 0 | 2
stomach pain (Gastrointestinal disorders) | 0 | 2
GERD (Gastrointestinal disorders) | 1 | 1
allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 | 0
bruising (Injury, poisoning and procedural complications) | 1 | 0
cardiac disorders (Cardiac disorders) | 0 | 1
chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
dehydration (Metabolism and nutrition disorders) | 0 | 1
dysphagia (Gastrointestinal disorders) | 1 | 0
ear pain (Ear and labyrinth disorders) | 1 | 0
diverticulitis (Gastrointestinal disorders) | 0 | 1
hemorroids (Gastrointestinal disorders) | 0 | 1
hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 | 1
menorrhagia (Reproductive system and breast disorders) | 0 | 1
pharyngitis (Infections and infestations) | 0 | 1
pregnancy, puerperium and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 0 | 1
presyncope (Nervous system disorders) | 1 | 0
rash (Skin and subcutaneous tissue disorders) | 0 | 1
renal and urinary disorders (Renal and urinary disorders) | 0 | 1
reproductive system and breast disorders (Reproductive system and breast disorders) | 0 | 1
sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
toothache (Gastrointestinal disorders) | 1 | 0
transient ischemic attack (Nervous system disorders) | 1 | 0
bladder tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ear and labyrinth disorders (Ear and labyrinth disorders) | 1 | 0
corneal ulcer (Eye disorders) | 0 | 1
infections and infestations (Infections and infestations) | 0 | 1
wound complication (Injury, poisoning and procedural complications) | 1 | 0
esophageal infection (Infections and infestations) | 1 | 0
lung infection (Infections and infestations) | 0 | 1
autoimmune disorder (Immune system disorders) | 0 | 1
dysuria (Renal and urinary disorders) | 1 | 0
noncardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
cystitis noninfective (Renal and urinary disorders) | 0 | 1
papularpustulo rash (Skin and subcutaneous tissue disorders) | 0 | 1
muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-07-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT01972308/Prot_SAP_000.pdf